CLINICAL TRIAL: NCT02704104
Title: A Randomized Controlled Single-Blind Investigation to Evaluate the Safety and Performance of the AC5 Topical Hemostatic Device (AC5™) Following Excision of Skin Lesions
Brief Title: Safety and Performance Evaluation of the Topical Hemostatic Device (AC5™) Following Excision of Skin Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arch Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AC5-1
Record Dates: First submitted 2016-03-01; First posted 2016-03-09 (Estimated); Results first posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Skin Neoplasms
Keywords: topical hemostat; self-assembling peptide barrier
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AC5 Topical Hemostatic Device (Experimental): The intervention in this arm is the application of a topical hemostatic agent (AC5) to a freshly excised skin lesion
  Interventions: Device: AC5 Topical Hemostatic Device
- Control (Placebo Comparator): The intervention in this arm is the application of saline (Control) to a freshly excised skin lesion
  Interventions: Device: AC5 Topical Hemostatic Device

INTERVENTIONS:
Device: AC5 Topical Hemostatic Device — Randomized application of the hemostatic agent AC5 to one of two freshly excised lesions in each patient

SUMMARY:
This study is designed to monitor patient safety after excision of skin lesions and subsequent application of AC5 topical hemostatic agent and to assess the performance of AC5 for controlling bleeding in skin wounds.

DETAILED DESCRIPTION:
This is a randomized, controlled single-blind pilot study to evaluate the safety and performance of AC5 following excision of lesions from the trunk or upper limbs under local anesthetic, in patients currently prescribed or not prescribed antiplatelet monotherapy.

Each patient had sequential shave excision of two lesions (one treatment, one Control) at the same sitting. The sequence of wound treatment (AC5 first or Control first) was randomized.

Study and Control treatments were administered immediately after lesion excision, followed by determination of time to hemostasis (TTH), and application of an occlusive water-resistant dressing

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18 and 85.
* Voluntary written informed consent, given before performance of any clinical investigation-related procedure not part of standard medical care, and with the understanding that consent may be withdrawn at any time without prejudice to future medical care.
* Scheduled for excision of 2 (two) or more skin lesions from their trunk or upper limbs (defined as lying below the level of the inferior border of the patient's mandible).
* If subjects is currently prescribed an antiplatelet therapy, it must from one of the following therapies at levels as per hospital protocol:
* Antiplatelet monotherapy with one of the following agents:

  * Aspirin
  * Clopidogrel (thienopyridine-class antiplatelet agent)
  * Ticagrelor
  * Dipyridamole
* Female subjects must meet at least one of the following additional criteria:

  * Surgically sterile with bilateral tubal ligation or hysterectomy.
  * Post-menopausal for at least one year.
  * If of child-bearing potential, practicing an acceptable method of birth control for the duration of the clinical investigation as judged by the Investigator, such as condoms, foams, jellies, diaphragm, intrauterine device or abstinence.
* Subjects willing to undergo pre-and post-clinical investigation blood and urine collection, physical exams and laboratory investigations.

Exclusion Criteria:

* Active infection as demonstrated by temperature > 37.5 C and clinical features of active infection.
* Wound expected to expose bone or tendon.
* Wound expected to require topical antibiotics.
* Know contraindication or reaction to Tegaderm use.
* Presence of malignancy or clinical expectation of malignancy based on examination.
* Known immunosuppression or taking immunosuppressive agents including systemic steroids.
* Plan for adjunctive flap or graft procedure to obtain closure of the wound(s) subject to this study.
* History of severe co-morbidity with expected patient survival ≤ 6 months.
* Pregnancy or lactation
* Intake of investigational drugs within 28 days prior to enrollment.
* Currently taking oral anticoagulants
* History of concurrent condition that, in the Investigator's opinion, would jeopardize the safety of the subject or compliance with the protocol.
* History of clinically significant, active disease (within 12 months prior to enrollment) of the pulmonary, gastrointestinal, neurological, genitourinary, renal, or haematological system, that in the opinion of the Principal Investigator, may confound the results of the trial or pose additional risk to the subject following the administration of AC5.
* History of clinically significant cardiac disorder, defined as: acute coronary syndrome, congestive heart failure (NYHA class III/IV), diagnosis of unstable angina pectoris, cerebral stroke and or myocardial infarction within the last 12 months or planned coronary or carotid revascularisation procedures anytime through 30 Day follow-up.
* History of severe uncontrolled treated or untreated hypertension (systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥100 mmHg).
* Likely inability to comply with the protocol or cooperate fully with the investigator and site personnel.
* Presence of significant cognitive impairment (Mini Mental Status Examination <22) or mental incapacity.
* Unwillingness or language barrier precluding adequate understanding of the trial procedure or cooperation with trial site personnel.
* Known or suspected active abuse of alcohol, narcotics or non-prescription drugs.
* Other planned surgical procedures within 30 days prior to or 30 days post-index procedure.
* Prior enrollment in this AC5 clinical trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack Kelly, MD, Principal Investigator — Professor of Surgery
Locations (1):
- University College Hospital, Galway, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wilson AP, Treasure T, Sturridge MF, Gruneberg RN. A scoring method (ASEPSIS) for postoperative wound infections for use in clinical trials of antibiotic prophylaxis. Lancet. 1986 Feb 8;1(8476):311-3. doi: 10.1016/s0140-6736(86)90838-x. PMID 2868173

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited who were to undergo excision of two skin lesions in the same sitting.
Groups:
- All Study Participants: All study participants had two freshly excised lesions, each randomized to either application of a topical hemostatic device (AC5) or control (saline) treatment.
Period: Overall Study
Arm/Group | All Study Participants
Started | 46
Completed | 46
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: Characteristics of the 46 patients enrolled in the study
Arm/Group | Overall
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 45
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Ireland | 46
Antiplatelet therapy [Count of Participants; unit: Participants] | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events Related to Clinical Investigation Product During the 30 Days of Follow-up
Description: Local reactions to clinical investigation product (pain, edema, rash, cellulitis, localized infectious processes, other) detected during clinical investigation follow up.
  Systemic reactions after administration of clinical investigation product (fever, allergic reaction, anaphylaxis or any clinical untoward event) detected during clinical investigation follow up.
Time Frame: 30 Days Post Procedure
Measure: Count of Participants; unit: Participants
Groups:
- AC5 Topical Hemostatic Device: The intervention in this arm is the randomized application of a topical hemostatic device (AC5) to one of two freshly excised lesions in each patient. Number in this arm refers to number of lesions
- Control: The intervention in this arm is the randomized application of saline (Control) to one of two freshly excised lesions in each patient. Number in this arm refers to lesions
Arm/Group | AC5 Topical Hemostatic Device | Control
Number analyzed (Participants) | 46 | 46
Participants | 2 | 3

2. Secondary Outcome: Median Time to Hemostasis (Seconds)
Description: Measure of time from application of treatment or control to the wound, to bleeding cessation
Time Frame: At time of application (Day 0)
Population: Analysis is performed per wound (2/patient, one randomized to AC5 the second to control), that is, 46 patients with a total of 96 wounds.
Measure: Median (Full Range); unit: seconds
Arm/Group | AC5 Topical Hemostatic Device | Control
Number analyzed (Participants) | 46 | 46
seconds | 24.5 [7 to 165] | 44 [10 to 387]

3. Secondary Outcome: Time to Hemostasis in Seconds Per Square Centimeter Wound Area
Description: Measure of time from application of treatment or control to the wound, to bleeding cessation/ divided by wound area
Time Frame: At time of application (Day 0)
Population: as for outcome 2
Measure: Median (Full Range); unit: seconds/cm2
Arm/Group | AC5 Topical Hemostatic Device | Control
Number analyzed (Participants) | 46 | 46
seconds/cm2 | 42 [5 to 1100] | 104 [6 to 797]

4. Secondary Outcome: Number of Wounds With ASEPSIS Wound Scores of 0 at Day 7 and Day 30
Description: The Additional treatment, the presence of Serous discharge, Erythema, Purulent exudate, and Separation of the deep tissues, the Isolation of bacteria, and the duration of inpatient Stay longer than 14 days (ASEPSIS) Wound Score (reference 1) was used to assess wound healing and overall wound sepsis. This multipoint system is reported as a total score ranging from 0 to 30 points in the first 7 days postoperatively. Additional points after 7 days can be added for additional treatments such as use of antibiotics, drainage of pus under local anesthesia, and debridement of the wound; and isolation of bacteria or duration of stay, for a total score of from 0 to 70 points by day 30. Total scores from 0-10 indicate satisfactory healing, from 11 to 20=disturbance of healing, from 21 to 30=minor wound infection, from 31 to 40=moderate wound infection, and >40 points signifies severe infection. For this study, the number of wounds with ASEPSIS score = 0 was counted.
Time Frame: 7 and 30 Days Post Procedure
Population: as for outcome 2
Measure: Number; unit: wounds
Groups:
- Wounds Treated With AC5 Topical Hemostatic Device: The intervention in this arm is the randomized application of a topical hemostatic device (AC5) to one of two freshly excised lesions in each patient. Number in this arm refers to number of wounds
- Wounds Treated With Control: The intervention in this arm is the randomized application of saline (Control) to one of two freshly excised lesions in each patient. Number in this arm refers to wounds
Arm/Group | Wounds Treated With AC5 Topical Hemostatic Device | Wounds Treated With Control
Number analyzed (Participants) | 46 | 46
wounds
  Day 7 | 40 | 40
  Day 30 | 44 | 44

5. Other Pre Specified Outcome: Time to Hemostasis in Patients Who Were Taking or Not Taking Anti Platelet Medication
Time Frame: Day 0
Population: The overall number of patients is 46, 10 of whom were taking anti platelet therapy at the time of the procedure.
Measure: Median (Full Range); unit: seconds
Arm/Group | AC5 Topical Hemostatic Device | Control
Number analyzed (Participants) | 46 | 46
seconds
  Taking antiplatelet therapy: number analyzed (Participants) | 10 | 10
  Taking antiplatelet therapy | 24 [7 to 120] | 90 [23 to 387]
  Not taking antiplatelet therapy: number analyzed (Participants) | 36 | 36
  Not taking antiplatelet therapy | 24 [8 to 165] | 40 [10 to 244]

ADVERSE EVENTS:
Time Frame: 30 days
Description: Adverse events were assessed immediately after treatment (Day 0), Day 7, and Day 30.
Groups:
- AC5 Topical Hemostatic Device: The intervention in this arm is the application of a topical hemostatic agent (AC5) to a freshly excised skin lesion
  AC5 Hemostatic agent: Randomized application of the hemostatic agent AC5 to one of two freshly excised lesions in each patient
- Control: The intervention in this arm is the application of saline (Control) to a freshly excised skin lesion
  AC5 Hemostatic agent: Randomized application of the hemostatic agent AC5 to one of two freshly excised lesions in each patient
Arm/Group | AC5 Topical Hemostatic Device | Control
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 13/46 | 13/46
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AC5 Topical Hemostatic Device (N=46) | Control (N=46)
Wound complication (Injury, poisoning and procedural complications) | 4 (5) | 4
Secretion discharge (General disorders) | 3 | 3
Fibrin D dimer increased (Investigations) | 2 | 2
Wound hemorrhage (Injury, poisoning and procedural complications) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No